CLINICAL TRIAL: NCT06973135
Title: Outcome Of Non-Surgical Single Visit Endodontic Retreatment in Teeth With Asymptomatic Apical Periodontitis Using Bioceramic Sealer (A Randomized Controlled Clinical Trial)
Brief Title: Non-Surgical Single Visit Endodontic Retreatment in Cases With Asymptomatic Apical Periodontitis Using Bioceramic Sealer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saly Nazeer (Other)
Responsible Party: Sponsor-Investigator, Saly Nazeer, doctor, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0966-09/2024
Record Dates: First submitted 2025-05-04; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Asymptomatic Apical Periodontitis; Root Canal Retreatment
Keywords: CBCT; secondary root canal treatment; asymptomatic apical periodontitis; bioceramic sealer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bioceramic sealer group (Active Comparator): obturation of mandibular molar root canals using bioceramic sealer after canal shaping and cleaning in single visit
  Interventions: Procedure: Bioceramic sealer root canal obturation
- resin sealer group (Active Comparator): mandibular molar root canal obturation using resin sealer after canal cleaning and shaping in single visit
  Interventions: Procedure: resin sealer root canal obturation

INTERVENTIONS:
Procedure: Bioceramic sealer root canal obturation — Mandibular molars root canal obturation with bioceramic sealer after non surgical endodontic retreatment and then immediate periapical radiograph will be done to record PAI
  Arms: bioceramic sealer group
Procedure: resin sealer root canal obturation — non surgical root canal retreatment of mandibular molar teeth will be done using resin based sealer in obturation and periapical radiograph will be taken immediately to record PAI
  Arms: resin sealer group

SUMMARY:
The goal of this clinical trial is to learn if using bioceramic sealers in non surgical single visit endodontic retreatment in patients with endodontic treatment failure and asymptomatic apical periodontitis will work in comparison to other resin sealer which proved efficacy ,and help healing of the periapical lesions and reduce the anticipated postoperative pain , Participants will have root canal retreatment done in a single visit and then follow up will be done in 1, 3 and 6 months to check healing and then after 12 months , also postoperative pain will be monitored through communicating the patients after 24, 28 , 72 hours and the 7 days

DETAILED DESCRIPTION:
selection of the cases will be done according to the eligibility criteria the a baseline periapical radiograph to record the periapical index and base line CBCT will be done to measure the lesion size and record the CBCTPAI then patients will be divided into two groups (A AND B) randomly to perform single visit non surgical root canal retreatment using bioceramic sealer in obturation in group A and resin sealer in group B then post operative pain assessment will be done using numerical scale after 24, 48, 72 hours and 7 days .for radiographical and clinical measuring of the healing follow up will done after 1, 3, 6 and 12 months by performing periapical radiographs and recording PAI and clinical signs or symptoms and CBCT after 12 months to record CBCTPAI and compare the size differences at baseline

ELIGIBILITY:
Inclusion Criteria:

1. Mandibular molar teeth with previous unsuccessful endodontic treatment from ≥ 1 year with asymptomatic apical periodontitis.
2. Teeth with inadequate obturation.
3. Teeth with broken instruments that can be bypassed and/or retrieved and not present in the apical third or passing through the apex.
4. Teeth with periapical lesion.
5. Patient with the ages of 18-65 years.
6. Patient medically healthy and free from systemic diseases or with mild controlled systemic disease. ASA I, II * (52).
7. Patient with no acute pain or extraoral swelling.
8. Patients who agreed to participate in the study and attend the control visits.

   -

Exclusion Criteria:

1. Teeth requiring retreatment with a poor prognosis (root canal morphology altered, large carious cavity, internal or external root resorption, root perforation)
2. Teeth with vertical root fracture or open apex.
3. Patient with systemic disorders related to bone metabolism and using drugs that may affect bone metabolism.
4. Pregnant patients.
5. Patient under antibiotics treatment 2 weeks before the treatment.
6. Patients who could not attend follow up will be excluded from the study

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Measure the healing of periapical lesions through comparing size of lesion using periapical radiograph and CBCT before and after 1 year follow up | 21 months
  periapical radiograph and cone beam computed tomography will be taken to measure the size of the lesion and record the PAI and CBCTPAI at baseline then root canal retreatment will be done in single visit using bioceramic sealer in obturation in group A and resin sealer in group B and then periapical radiograph will be taken after 1, 3, 6 , 12 months to record PAI and CBCT at 12 months to record CBCTPAI to evaluate healing through measuring the sizes of periapical lesions , together with clinical record of the patients symptoms after 1, 3 ,6 and 12 months

SECONDARY OUTCOMES:
Clinical assessment of post operative pain | 21 months
  The postoperative pain will be recorded using a numeric rating scale (NRS) on a 0-10 scale, with 0 indicating no pain and 10 indicating the worst pain. Patients were required to report their pain level at 4-time intervals after obturation: 24, 48, 72 hours and 7 days. The highest pain score recorded at 3 consecutive time points will be selected

CONTACTS AND LOCATIONS:
Overall Officials: Sybel M Moussa, Phd, Study Director — Alexandria University; Nehal Lehita, Phd, Study Director — Alexandria University
Locations (1):
- faculty of dentistry Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study design and statistical analysis
Supporting Information: SAP
Time Frame: from January 2025 with no end date
Access Criteria: study protocol and other data relative to the study is available at Alexandria university faculty of dentistry official site , can be accessed by anyone who would ask for
URL: https://dent.alexu.edu.eg/index.php/ar/

REFERENCES:
- Available data/document: Statistical Analysis Plan — https://dent.alexu.edu.eg/index.php/ar/

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT06973135/SAP_000.pdf